CLINICAL TRIAL: NCT02558244
Title: Impact of Image-defined Risk Factors on the Outcome of Patients With Neuroblastoma: A Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Morsy, MD, Lecturer, Pediatric Oncology Department, Assiut University
Other Study IDs: Image-defined RF NB
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Neuroblastoma
Keywords: Childhood Cancer; Image-defined Risk Factors; Pediatric Oncology
MeSH Terms: conditions — Neuroblastoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate Image-defined Risk Factors (IDRF) in patients with neuroblastoma, at the time of their initial presentation, as a prognostic factor for prediction of subsequent outcome & complications related to surgery, in the accordance with the experience of South Egypt Cancer Institute (SECI), which is the largest referral site in Upper Egypt.

DETAILED DESCRIPTION:
Background:

Neuroblastoma is the third most common childhood cancer, after leukemia and brain tumors, and is the most common solid extracranial tumor in children.

The concept of surgical risk factors in neuroblastoma surgery was introduced with the European multicenter study (LNESG1) study.

In 2005 the International Neuroblastoma Risk Group (INRG) Task Force, representing all major co-operative pediatric cancer groups, adopted the principle of surgical risk factors and incorporated it in the INRG Staging System. The INRG Task Force preferred the term Image-Defined Risk Factors (IDRF) to surgical risk factors, and agreed upon a list of IDRF.

Patients & Methods:

This retrospective study will be carried out by reviewing the medical records of patients with neuroblastoma seen at the pediatric oncology department, in the period from 2001 January till 2015 December.

Data from Patients' medical records will be gathered, Pathologic diagnosis of neuroblastoma will be verified before the enrollment into the study. As an initial imaging was done for all patients at presentation, as a routine for diagnosis & staging, the reports of the computed tomography scans will be reviewed for verification of the presence or absence of the IDRF. This historical cohort will be followed forward with time for ascertainment of the role of surgery in treatment, and treatment outcomes of these patients. Any complications occurred due to surgery will be reported, as collected from surgical reports of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age less than 19 years.
* Patients diagnosed with non-metastatic neruoblastoma.

Exclusion Criteria:

* Patients whose age more than 18 years.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cancer patients, those diagnosed with Neuroblastoma, in the period from 2001 January till 2015 December, and received treatment at the pediatric oncology department, their medical records will be retrospectively reviewed for data collection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Participants will be retrospectively followed forward in time from the date of diagnosis till the primary completion date of the study, an expected average of 5 years
  Time from the date of diagnosis until death from any cause
Event Free Survival (EFS) | Participants will be retrospectively followed forward in time from the date of diagnosis till the primary completion date of the study, an expected average of 5 years
  Time from the date of diagnosis until disease progression, or death for any reason.

SECONDARY OUTCOMES:
Complications of Surgery | Participants will be retrospectively followed forward in time from the date of surgical operation till the occurence of any complication due to surgery, an expected average of 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Cecchetto G, Mosseri V, De Bernardi B, Helardot P, Monclair T, Costa E, Horcher E, Neuenschwander S, Toma P, Rizzo A, Michon J, Holmes K. Surgical risk factors in primary surgery for localized neuroblastoma: the LNESG1 study of the European International Society of Pediatric Oncology Neuroblastoma Group. J Clin Oncol. 2005 Nov 20;23(33):8483-9. doi: 10.1200/JCO.2005.02.4661. PMID 16293878
- [Background] Monclair T, Brodeur GM, Ambros PF, Brisse HJ, Cecchetto G, Holmes K, Kaneko M, London WB, Matthay KK, Nuchtern JG, von Schweinitz D, Simon T, Cohn SL, Pearson AD; INRG Task Force. The International Neuroblastoma Risk Group (INRG) staging system: an INRG Task Force report. J Clin Oncol. 2009 Jan 10;27(2):298-303. doi: 10.1200/JCO.2008.16.6876. Epub 2008 Dec 1. PMID 19047290
- [Background] Brisse HJ, McCarville MB, Granata C, Krug KB, Wootton-Gorges SL, Kanegawa K, Giammarile F, Schmidt M, Shulkin BL, Matthay KK, Lewington VJ, Sarnacki S, Hero B, Kaneko M, London WB, Pearson AD, Cohn SL, Monclair T; International Neuroblastoma Risk Group Project. Guidelines for imaging and staging of neuroblastic tumors: consensus report from the International Neuroblastoma Risk Group Project. Radiology. 2011 Oct;261(1):243-57. doi: 10.1148/radiol.11101352. Epub 2011 May 17. PMID 21586679